CLINICAL TRIAL: NCT04717674
Title: An Investigation of Short-chain Fatty Acid Uptake in Solid Tumours as Assessed by [18F]Fluoropivalate Positron Emission Tomography and Its Relationship With Tumour Proliferation
Brief Title: [18F]FPIA PET/CT Imaging in Patients With Solid Tumours
Acronym: [18F]FPIA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); Imperial College London (Other); National Cancer Imaging Translational Accelerator (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 135083
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Tumor, Solid
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug: [18F]Fluoropivalate ([18F]Fluoro-2,2-Dimethylpropionic Acid) (FPIA) (Experimental): Participants will undergo two PET/CT scans with the tracer [18F]Fluoropivalate ([18F]Fluoro-2,2-Dimethylpropionic Acid) (FPIA), referred to as [18F]FPIA, on 2 separate visits.
  Interventions: Drug: [18F]Fluoropivalate ([18F]Fluoro-2,2-Dimethylpropionic Acid); Procedure: PET/CT

INTERVENTIONS:
Drug: [18F]Fluoropivalate ([18F]Fluoro-2,2-Dimethylpropionic Acid) — [18F]FPIA radiotracer administration
  Other Names: None are used.
Procedure: PET/CT — PET/CT scan

SUMMARY:
The study will be a phase 2, open-label study in patients with solid tumours to explore the relationship between short-chain fatty acid uptake using [18F]FPIA PET/CT and tumour proliferation

DETAILED DESCRIPTION:
Cancers have increased energy demands to allow for their rapid growth compared to healthy cells. Glucose is the main source of energy for many cells in the body, and clinicians routinely use a scan which looks at glucose metabolism to assess if cancer treatment is working. However, some cancer cells can create energy to survive and grow in a different way, using fatty acids. In this study, the investigators are using a PET/CT scan to look at a variety of cancer types to see which cancers use fatty acids for energy and if this can be measured. The PET/CT scan will be carried out twice on 2 separate visits so that the investigators can check that both scans give the same result.

The investigators will also carry out special tests on the tumour tissue taken during routine cancer surgery. These tests will look for specific substances in the cancer cells that are related to cancer biology and growth. The investigators will then compare the results from the surgical tissue to the results of the scan to see if there is a relationship between them.

The study will look at 21 patients with solid tumours conducted in 4 NCITA accredited centres, which have different strengths in recruiting specific patient/tumour-type cohorts. Each patient will have two scan visits (between 2-15 days apart) prior to any new treatment starting to check that the scan measurements are repeatable.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiological evidence of solid primary or metastatic target tumour lesions and the following characteristics will be recruited:

  1. Age ≥18 years of age
  2. Radiologically confirmed tumour size ≥15mm (at least one lesion must be extra-hepatic)
  3. The participant is due to undergo surgery within 3 months of the first [18F]FPIA PET/CT
  4. There is time to complete the two research PET studies without any delay to surgery
  5. WHO performance status 0 -2
  6. If female, the participant is either post-menopausal (>1 year), or surgically sterilised (has had a documented bilateral oophorectomy and/or documented hysterectomy, >2 years), or if of childbearing potential, must have a negative urine pregnancy test within 2 hours prior to injection of imaging agent
  7. The participant is able and willing to comply with study procedures, and signed and dated informed consent is obtained.
  8. eGFR of ≥30 within 3 months of [18F]FPIA injection.
  9. The participant is not scheduled to start cancer treatment (e.g. chemotherapy, radiotherapy, biological therapy or immunotherapy) within the study scanning period.

Exclusion Criteria:

* 1. The participant has received chemotherapy, immunotherapy, biologic therapy or investigational therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of [18F]FPIA injection or is due neoadjuvant therapy between the PET and surgery.

  2. The participant is pregnant or lactating. 3. The participant is scheduled to have a nuclear medicine or contrast scan within 24 hours before the administration of [18F]FPIA.

  4. Participants with claustrophobia or who are unable to comfortably tolerate the scanning procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The relationship between [18F]FPIA uptake and percent positive tumour cells reported as counts defined per area from whole section immunohistochemistry for PHH3. | 6 months
  To explore the relationship between short-chain fatty acid uptake using [18F]FPIA PET/CT and tumour proliferation in patients with solid tumours.

SECONDARY OUTCOMES:
Estimation of SUVmax of target lesions at 30 minutes and 60 min. | 60 min
  The SUVmax of the target lesions will be estimated for both timepoints (i.e. 30 min and 60 min) in order to assess changes in this measurand at the two time points.
Estimation of tumour-to-background ratio of target lesions at 30 minutes and 60 min. | 60 min
  The tumour-to-background ratio of the target lesions will be estimated for both timepoints (i.e. 30 min and 60 min), in order to assess changes in this measurand at the two time points.
Graphical presentation and reliability of repeat semi-quantitative measure (SUV) of target lesions between two PET scans for each time point (30 min and 60 min). Bland Altman and ICC will be presented. | 15 days
  To assess the repeatability of the two [18F]FPIA PET scans, as this can impact the primary end point. The two [18F]FPIA PET scans will be 2-15 days apart, and each will consist of two imaging timepoints (30 minutes and 60 minutes).
Graphical presentation of [18F]FPIA uptake and whole section immunohistochemistry for Ki-67 and mitotic count (mitoses per mm2) assessed on hematoxylin and eosin (H&E) sections. Pearson's correlation coefficient will be reported. | 6 months
  To explore the relationship between [18F]FPIA PET/CT and other known tumour proliferation markers

OTHER OUTCOMES:
To explore the relationship between [18F]FPIA tumour uptake and histological markers of tumour metabolism. | 6 months
  Graphical and tabular description of the relationship of [18F]FPIA uptake with biological markers including pan-mitochondrial markers (succinate dehydrogenase [SDHA], citrate synthase), and fatty acid oxidation enzymes (carnitine palmitoyltransferase I/carnitine acyltransferase I [CPT1/CAT1], carnitine-acylcarnitine translocase [CACT], SLC22A2, SLC22A5, and SLC25A20), evaluated by IHC

CONTACTS AND LOCATIONS:
Overall Officials: Tara Barwick, Principal Investigator — University College, London
Locations (3):
- United Kingdom (3):
  - Guy's & St. Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, London